CLINICAL TRIAL: NCT06965686
Title: Development of a Personalized, Psychosocial Intervention for Menopausal Individuals With Elevated Dementia Risk
Acronym: PERI-MIND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB24-1148
Record Dates: First submitted 2025-04-15; First posted 2025-05-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Menopausal; Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perimenopausal individuals with a family history of dementia (Experimental): For the focus groups, the investigators will recruit a minimum of 20 participants. Participants will take part in a single 1-hour remote focus group session, where they will be asked about their fears about dementia, informational and decisional needs, and strategies to promote adaptive coping as they transition through menopause.
  For pilot testing, we will recruit a minimum of 30 participants. Participants will be asked to evaluate the online intervention materials across 3-weeks. The evaluation will focus on feasibility and acceptability of the intervention.
  Interventions: Behavioral: PERI-MIND

INTERVENTIONS:
Behavioral: PERI-MIND — PERI-MIND will be informed by the focus group findings from phase one. However, the investigators anticipate including core components related to psychoeducation, psychological grounding, & behavioral activation, which will be specifically adapted to the perimenopausal and menopausal population. Psychoeducation in this context will focus on menopausal symptoms like brain fog (e.g., how common they are, how long they typically last), information about dementia and its risk factors (e.g., most actionable risk factors in mid-life), and links between menopause and dementia (e.g., hormonal replacement therapy). Psychological grounding content will focus on practical training exercises in mindful monitoring of concerns about brain fog and other menopausal symptoms (e.g., meditation, deep breathing). Behavioral activation will focus on exercises to recognize and disrupt avoidant coping behaviors, and increase engagement in valued activities (e.g., social engagement, exercise, healthy eating).

SUMMARY:
By age 45, women's lifetime risk of dementia is estimated to be 1 in 5. Two-thirds of people currently living with a dementia diagnosis are women, and-women make up the majority of carers for people with dementia. Because women bear a larger burden of the dementia epidemic, they tend to be more fearful about dementia compared to men. Women may be especially fearful during the menopause transition, which can impact cognition. These fears can cause significant psychological distress, functional impairment, and avoidance of help seeking. Interventions that acknowledge women's fears and promote adaptive coping during the menopause transition are needed to combat dementia-related fear and its negative impacts.

This project aims to develop, and pilot test a brief personalized, psychosocial intervention for middle-aged perimenopausal individuals with elevated dementia risk. The investigators will assess the intervention's acceptability and feasibility for use in this population. The project will be completed in three stages. First, the investigators will conduct focus groups to better understand individual fears about dementia, informational and decisional needs, and strategies to promote adaptive coping as they transition through menopause (case-only, single time point). Second, the investigators will develop an intervention to meet the specific needs identified by the focus groups. Intervention components will address multiple areas of women's health in midlife, including aspects of physical and psychological health, as well as functional health outcomes that have important and long-lasting life implications. Finally, the investigators will conduct pilot testing to assess the acceptability and feasibility of the intervention (cohort, 3-week testing period).

This project will deliver a novel psychosocial intervention that can provide middle-aged perimenopausal women with the information and practical skills that can help them manage their dementia-related fears and encourage adaptive coping behaviors. Outputs from the project will serve as preliminary data for a fully powered randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Female sex at birth
* Aged between 40-58 years
* Late perimenopause or early post-menopause
* Elevated dementia risk characterized by first degree relative with diagnosis of Alzheimer's disease or another dementia

Exclusion Criteria:

* Diagnosis of Mild Cognitive Impairment, Alzheimer's or another dementia
* Diagnosis of other chronic illness or condition that affects cognition (e.g., Axis I psychiatric disorders such as schizophrenia or mood disorders, neurological disorders such as stroke, cancer, traumatic brain injury)
* Inadequate vision or hearing to engage with intervention materials
* Unable or unwilling to provide informed consent
* Iatrogenic menopause (i.e., due to surgery)

Ages: 40 Years to 58 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who are enrolled and complete the study | From enrollment until pilot testing is completed
  Feasibility outcomes will relate to the successful implementation and completion of the intervention, including the ease of recruitment and ability of participants to enroll and complete the study. Metrics will include the total number of participants identified and enrolled in the study and completion rate.
Acceptability of intervention content | From enrollment until pilot testing is completed
  Acceptability will be assessed using standard Likert-type scales, informed by the Theoretical Framework of Acceptability for healthcare interventions. Questions will focus on the content, presentation format and length.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Farina, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets generated and analyzed during the study will be made available in the Open Science Framework (OSF) repository on completion of the study: https://osf.io/cwn79/.
Time Frame: IPD and supporting information will be made permanently available online on completion of the study.
Access Criteria: De-identified data will be made available to researchers, the public and funders.
URL: https://osf.io/cwn79/

REFERENCES:
- See also: Related Info — https://obgyn.uchicago.edu/research/peri-mind